CLINICAL TRIAL: NCT03886779
Title: Clinical Outcomes of Prolensa (Bromfenac Ophthalmic Solution) 0.07% QD vs. Ilevro (Nepafenac Ophthalmic Suspension) 0.3% QD With Extra (Pulse) Dose on Day of Surgery for Treatment of Ocular Inflammation Associated With Cataract Surgery in a Randomized, Single Masked Clinical Trial
Brief Title: Study Title: Clinical Outcomes of Prolensa (Bromfenac Ophthalmic Solution) 0.07% QD vs. Ilevro (Nepafenac Ophthalmic Suspension) 0.3% QD With Extra (Pulse) Dose on Day of Surgery for Treatment of Ocular Inflammation Associated With Cataract Surgery in a Randomized, Single Masked Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Silverstein Eye Centers (Other)
Collaborators: Bausch & Lomb Incorporated (Industry); Churchhill Communications (Unknown); Statistics & Data Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLMAIIT-02-13
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Treatment of Ocular Inflammation Associated With Cataract Surgery
Keywords: Post-Ocular Inflammation; Cataract Surgery
MeSH Terms: interventions — bromfenac; nepafenac

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, investigator masked, parallel group, and active-comparator controlled study to evaluate the clinical outcomes of Prolensa (Bromfenac Ophthalmic Solution) 0.07% for the treatment of ocular inflammation associated with cataract surgery
Who Masked: Investigator
Masking Description: The study is investigator-masked to treatment group assignment for the duration of the study.
  Should the masking need to be broken, the study staff may reveal the treatment to the Investigator. The date, time, and reason for the unmasking must be documented as soon as
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prolensa (Bromfenac Ophthalmic Solution) 0.07% (Active Comparator): Bausch and Lomb, Rochester, NJ Dose: Subjects will instill one drop into the study (operative) eye once daily for a maximum of 16 days. Dosing will begin one days prior to surgery (Day 1), continue on the day of surgery plus 1 hour before surgery and for 14 days after surgery.
  Interventions: Drug: Bromfenac
- Ilevro® (nepafenac ophthalmic suspension ) 0.3% (Active Comparator): Alcon Laboratories, Inc., Fort Worth, TX Dose: Subjects will instill one drop of test article into the study (operative) eye once daily for a maximum of 16 days. Dosing will begin one day prior to surgery (Day 1), continue on the day of surgery plus1 hour before surgery and for 14 days after surgery.
  Interventions: Drug: Nepafenac

INTERVENTIONS:
Drug: Bromfenac — 0.7 MG/ML [Prolensa]
  Arms: Prolensa (Bromfenac Ophthalmic Solution) 0.07%
Drug: Nepafenac — 3 MG/ML [Ilevro]
  Arms: Ilevro® (nepafenac ophthalmic suspension ) 0.3%

SUMMARY:
Clinical Outcomes of Prolensa (Bromfenac Ophthalmic Solution) 0.07% QD vs. Ilevro (nepafenac Ophthalmic Suspension) 0.3% QD with extra (pulse) dose on day of surgery for Treatment of Ocular Inflammation Associated with Cataract Surgery

DETAILED DESCRIPTION:
Name of Finished Product:

Prolensa (Bromfenac Ophthalmic Solution) 0.07% Bausch and Lomb, Rochester, NJ Dose: Subjects will instill one drop into the study (operative) eye once daily for a maximum of 16 days. Dosing will begin one days prior to surgery (Day 1), continue on the day of surgery plus 1 hour before surgery and for 14 days after surgery.

2) Ilevro® (nepafenac ophthalmic suspension ) 0.3% This is a single-center, randomized, investigator and subject-masked, parallel group, and active-comparator controlled study.

Subjects will be screened for this study between 1 and 21 days prior to the initiation of dosing with the test article. Subjects who sign the informed consent form and meet all inclusion/exclusion criteria will be randomized to receive either Prolensa (Bromfenac Ophthalmic Solution) 0.07% QD or Ilevro (nepafenac Ophthalmic Suspension) 0.3% (1:1) for 14 days after cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female at least 18 years of age who are scheduled for unilateral cataract surgery VIA phacoemulsification with posterior chamber intraocular lens implantation and for whom no other ophthalmic surgical procedures (e.g., relaxing incisions, iridectomy, conjunctival excisions, etc) are to be conducted during the cataract surgery.
2. Agree not to have any other ocular surgical procedures in the study or fellow (non study) eye within 15 days prior to the initiation of dosing with the test article or throughout the duration of the study.
3. Have a Best Corrected Visual Acuity of 20/200 or better in either eye.
4. Are willing/able to return for all required study visits.
5. Are willing/able to follow instructions from the study investigator and his/her staff.
6. Are able to self administer test article (or have a caregiver available to instill all doses of test article).
7. If a woman capable of becoming pregnant, agree to have urine pregnancy testing performed at screening (must be negative) and agree to use a medically acceptable form of birth control throughout the study duration and for at least one week prior to and after completion of the study. Women considered capable of becoming pregnant include all females who have experienced menarche and who have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
8. Have signed informed consent approved by Institutional Review Board or Independent Ethics Committee.
9. Have IOP ≥ 5 mmHg and ≤ 22 mmHg (in study eye) without anti glaucoma therapy at the pre operative screening visit (if >22 mmHg, adjust following pachymetry)

Exclusion Criteria:

1. Have known hypersensitivity to bromfenac or nepafenac or to any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
2. Have a known hypersensitivity to salicylates (i.e., aspirin) or to other non steroidal anti inflammatory drugs (NSAIDs).
3. Have intraocular inflammation (i.e., cells or flare in the anterior chamber as measured on slit lamp examination) in the study eye at the screening visit.
4. Have a known blood dyscrasia or bone marrow suppression, a diagnosis of uncontrolled/unstable peptic ulcer disease, inflammatory bowel disease, or ulcerative colitis, or any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease.
5. Have used ocular, topical, or systemic NSAIDs or ocular, topical, or systemic gentamicin, or cyclosporine ophthalmic emulsion within 7 days prior to initiation of dosing with the test article or throughout the duration of the study.
6. Have used any ocular prostaglandins within 30 days prior to initiation of dosing with the test article or throughout the duration of the study.
7. Have active corneal pathology noted in the study eye at the screening visit. Active corneal pathology is defined as corneal pathology that is non stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment. Superficial punctate keratitis in the study eye is a criterion for exclusion.
8. Have any extraocular/intraocular inflammation in the study eye noted at the screening visit (blepharitis allowed if mild only, and no concurrent conjunctivitis or lid erythema/edema) or ongoing, unresolved uveitis.
9. Have used topical, ocular, inhaled or systemic steroids within 14 days prior to screening.
10. Have had radial keratotomy, corneal transplant, or corneal refractive surgery in the study eye within the last two years.
11. Have a history of abuse of alcohol/drugs within six months prior to the screening visit.
12. Are pregnant or nursing/lactating.
13. Have participated in any other study of an investigational drug or device within 30 days prior to randomization.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Outcome Change measured by Summed Ocular Inflammation Score (SOIS) | Day 1 through Day 15
  50 Subjects are planned, 25 per treatment group who are undergoing planned cataract extraction with posterior chamber intraocular lens implantation to evaluate the non-inferiority of Prolensa and Ilevro when administering a pulse dose in each arm 1 hour prior to surgery. Outcome measure is defined as SIOS score of zero (no cell or flare) on day 15 (day one being the day prior to surgery, and for 14 days following surgery

SECONDARY OUTCOMES:
Adverse Events | 42 Days
  Adverse Events reported, elicited, and observed
Slit Lamp Biomicroscopy | 42 Days
  Slit Lamp Biomicroscopy evaluated and observed within normal limits
Intraocular Pressure | 42 Days
  Intraocular Pressure evaluated and observed within normal limits
Funduscopic Examination (Dilated) | 42 Days
  Funduscopic Examination (Dilated) evaluated and observed within normal limits

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Silverstein, MD, Principal Investigator — Silverstein Eye Centers

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: To Be Determined

REFERENCES:
- [Derived] Silverstein SM. Bromfenac Ophthalmic Solution 0.07% Versus Nepafenac Ophthalmic Suspension 0.3% for Post-Cataract Surgery Inflammation: A Pilot Study of Identical Dosing Regimens with Pre-Surgical "Pulse" Dose. Ophthalmol Ther. 2019 Dec;8(4):577-587. doi: 10.1007/s40123-019-00215-y. Epub 2019 Sep 24. PMID 31552543